CLINICAL TRIAL: NCT01541709
Title: A Phase II Study of Imatinib Dose Escalation to 800 mg/Day in Korean Patients With Metastatic or Unresectable GIST Harboring KIT Exon 9 Mutation: Imatinib Dose Escalation
Brief Title: Imatinib Dose Escalation to 800 mg/Day in Korean Patients With Metastatic or Unresectable GIST Harboring KIT Exon 9 Mutation: KENEDI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Min-Hee Ryu, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC1102
Record Dates: First submitted 2012-02-24; First posted 2012-03-01 (Estimated); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: This is a single-center; prospective; single-arm; open-label phase II study
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Imatinib (Experimental)
  Interventions: Drug: imatinib

INTERVENTIONS:
Drug: imatinib — The patients will receive 400 mg per day of imatinib for 4 weeks, and then 600mg per day (300 mg po bid) for 4 weeks if tolerable to 400 mg per day, and then 800 mg per day (400 mg po bid)

SUMMARY:
KIT exon 9 mutants had poorer survival compared with KIT exon 11 mutants when they were treated with the same dose of imatinib, 400 mg per day, and that patients with KIT exon 9 mutation had better progression-free survival with imatinib treatment at an escalated dose, 800 mg per day, than with imatinib treatment at a dose of 400 mg per day.10,11 Based on the results, imatinib 800 mg per day is now considered the standard dose for the treatment of patients with metastatic or unresectable GIST showing KIT exon 9 mutation in Western countries.

DETAILED DESCRIPTION:
According to our previous prospective phase II study of imatinib 400 mg per day in metastatic or unresectable GIST, hematologic and non-hematologic toxicities were more frequent in Korean patients compared to the Western studies.7 It may be caused by relatively higher exposure to imatinib per body surface area in Korean patients than in Western population because the weight and height of Korean patients are relatively smaller than Western people. So, we plan to start imatinib at 400 mg per day and then sequentially escalate the doses of imatinib in this study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Histologically confirmed metastatic or unresectable GIST with CD117(+), DOG-1 (+), or KIT mutation
* ECOG PS(Eastern Cooperative Oncology Group Performance Status) 0~2
* Primary mutation at KIT exon 9
* Imatinib treatment for less than 4 weeks from the first dose at 400 mg per day
* No prior use of tyrosine kinase inhibitors ((but, patients who have recurrence 6 months after completion of adjuvant imatinib at a dose of 400 mg per day can be enrolled in this study)
* At least one evaluable disease by RECIST v1.0
* Resolution of all toxic effects of prior treatments (chemotherapy, surgery, RFA(radiofrequency ablation), radiotherapy, and/or TACE)
* Adequate bone marrow function as defined by platelets ≥ 75 x 109/L and neutrophils ≥ 1.5 x 109/L (within 1 week prior to the first dose of imatinib at 400 mg per day)
* Adequate renal function, with serum creatinine < 1.5 x ULN (within 1 week prior to the first dose of imatinib at 400 mg per day)
* Adequate hepatic function with serum total bilirubin < 1.5 x ULN, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 2.5 x ULN in the absence of liver metastases, or < 5 x UNL in the presence of liver metastases (within 1 week prior to the first dose of imatinib at 400 mg per day)
* No other malignant disease apart from non-melanotic skin cancer or carcinoma in situ of the uterine cervix or any other cancer except where treated with curative intent > 5 years previously without evidence of relapse
* Provision of a signed written informed consent

Exclusion Criteria:

* Severe co-morbid illness and/or active infections
* Pregnant or lactating women
* History of other malignancies except basal cell carcinoma and carcinoma in situ of uterine cervix
* CNS metastasis
* Clinically significant bleeding in GI tract
* GI obstruction or malabsorption
* Known hypersensitivity to imatinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | up to 24months
  evaluated with Triphasic or dynamic CT scans of abdomen & pelvis, and other involved sites. Follow-up CT scans will be performed at 4 weeks and 12 weeks after the first dose of imatinib at 400 mg per day, and then every 3 months until disease using RECIST(Response Evaluation Criteria in Solid Tumors) version 1.0

SECONDARY OUTCOMES:
disease control rate | Up to 24weeks
safety control rate | up to 24months
overall survival (OS) | up to 24months
imatinib PK(pharmacokinetics) (Cmin) | up to 24months
percentage of successful dose escalation | up to 24months

CONTACTS AND LOCATIONS:
Overall Officials: Min-Hee Ryu, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, South Korea